CLINICAL TRIAL: NCT03117257
Title: A Prospective Phase II Randomized Clinical Trial: Docetaxel and Loplatin Induction Chemotherapy Followed by Concurrent Lobaplatin Chemoradiotherapy for Locally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: Docetaxel and Loplatin Induction Chemotherapy Followed by Concurrent Chemoradiotherapy for Locally Advanced SCCHN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guiyang Medical University (Other)
Responsible Party: Principal Investigator, Feng Jing, Head and neck cancer director, chief researcher, clinical professor, Guiyang Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20160819
Record Dates: First submitted 2017-04-02; First posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Locally Advanced Head and Neck Squamous Cell Carcinoma
Keywords: Lobaplatin; head and neck cancer; chronic-chemotherapy
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — lobaplatin; Platinum; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the treatment group (Experimental): docetaxel plus lobaplatin induction chemotherapy combined with lopoplatin chemoradiotherapy
  Interventions: Drug: Lobaplatin
- the control group (Active Comparator): TPF induction chemotherapy combined with cisplatin chemoradiotherapy
  Interventions: Drug: Cisplatin

INTERVENTIONS:
Drug: Lobaplatin — Device: Chrono-chemotherapy Drug: induction Chrono-chemotherapy Drug: Lobaplatin chrono-chemotherapy Radiation: intensity-modulated radiation therapy
  Other Names: Platinum
  Arms: the treatment group
Drug: Cisplatin — Device: Chrono-chemotherapy Drug: induction Chrono-chemotherapy Drug: cisplatin chrono-chemotherapy Radiation: intensity-modulated radiation therapy
  Other Names: cis-DDP; cis-Diammineplatinum(II) dichloride;
  Arms: the control group

SUMMARY:
This study is to observe and compare the safety and tolerability of docetaxel plus lobaplatin induction chemotherapy combined with lopoplatin chemoradiotherapy and TPF induction chemotherapy combined with cisplatin chemoradiotherapy in the treatment of locally advanced head and neck squamous cell carcinoma.

DETAILED DESCRIPTION:
TPF program is currently the local advanced head and neck squamous cell carcinoma commonly used inducing chemotherapy, cisplatin is the preferred drug for the same period chemotherapy, however, due to heavier gastrointestinal reactions caused by cisplatin， direct damage to renal parenchymal and other adverse reactions often lead to anti-tumor therapy can not be smooth Carried out, resulting in treatment failure, thus affecting the survival of patients. Therefore, how to improve the efficacy of the same time to reduce adverse drug reactions, as a prominent problem. Lobaplatin as the third generation of platinum antitumor drugs, anti-cancer activity and cisplatin rather, more than carboplatin. In this study, Phase II clinical trials were performed. Patients with locally advanced head and neck squamous cell carcinoma were randomly divided into experimental group and control group. The trial group was treated with docetaxel + lorosine-induced chemotherapy combined with lorplatin concurrent radiotherapy and chemotherapy. The control group was treated with TPF Cisplatin concurrent chemotherapy, observed and compared the efficacy and toxicity of the two treatment to assess its safety and patient tolerance.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation and written informed consent
2. Age 18-70 years old, gender is not limited
3. histologically proved to be squamous cell carcinoma
4. No surgery: head and neck squamous cell carcinoma 2010UICC staging Ⅲ - ⅣA, ⅣB period.

   After surgery: 2010UICC staging ⅣA, ⅣB;stage III tongue base or hypopharyngeal primaries;Postoperative naked eye or image residual stage III patients
5. Karnofsky score ≥70
6. Survival is expected to be ≥ 6 months
7. Women of childbearing age should be guaranteed contraception during the study period
8. (WBC) ≥4 × 109 / L * (unit normal), platelet (PLT) ≥100 × 109 / L (unit normal value), neutrophil cell (WBC), hematocrit (WBC) ≥1.5 × 109 / L * (unit normal value)
9. liver function: alanine aminotransferase (ALAT), aspartate aminotransferase (ASAT) <upper limit of normal (ULN) 1.5 times; total bilirubin <1.5 × ULN
10. renal function: serum creatinine <1.5 × ULN, endogenous creatinine clearance rate (Ccr) ≥ 55 ml / min
11. no serious complications such as hypertension, diabetes, coronary heart disease and psychiatric history
12. The treatment for the first course of treatment (no head and neck radiotherapy, no chemotherapy within 3 months).

Exclusion Criteria:

1. There is a distant shift
2. primary lesions or lymph nodes were radiotherapy
3. had received epidermal growth factor targeted therapy
4. primary tumor had received chemotherapy or immunotherapy
5. had other malignancies (except for cured basal cell carcinoma or cervical cancer)
6. pregnant women or lactating women and treatment during the observation period of contraceptive women of childbearing age
7. have a serious history of allergies or specific physical
8. Abuse of drugs or alcohol addicts
9. Person who has personality or mental illness, no civil capacity or limited civil capacity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2016-08-19 (Actual); Primary Completion 2019-08-19 (Estimated); Study Completion 2021-08-20 (Estimated)

PRIMARY OUTCOMES:
National Cancer Institute CTCAE v4.0 | 1 year
  Acute toxicity of radiotherapy and chemotherapy
evaluation of immediate efficacy | 1 year
  Evaluation of efficacy by RESIST1.1 standard

SECONDARY OUTCOMES:
overall survival | 5 years
  Evaluate the Overall survival at five years after Concurrent chemo-radiotherapy by RECIST.
progression-free survival | 5 years
  Evaluate the Progression-free survival at five years after Concurrent chemo-radiotherapy by RECIST.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Jin, Bachelor, Study Chair — Guizhou Provincial Cancer Hospital
Locations (1):
- Cancer Hospital of Guizhou Medical University, Guiyang, Guizhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang M, Chen Y, Wu W, Jin F, Li Y, Long J, Luo X, Gong X, Chen X, Liu L, Tang H, Wang Z. A prospective phase II randomized study of docetaxel combined with lobaplatin versus TPF regimen induction chemotherapy followed by concurrent chemoradiotherapy for locally advanced head and neck squamous cell carcinoma. J Cancer Res Clin Oncol. 2023 Dec;149(20):18081-18091. doi: 10.1007/s00432-023-05497-1. Epub 2023 Nov 20. PMID 37985501